CLINICAL TRIAL: NCT03838341
Title: Stand-Alone Thoracoscopic Epicardial Left Atrial Appendage Occlusion With AtriClip® Device for Thromboembolism Prevention in Nonvalvular Atrial Fibrillation - the Polish Nationwide Registry.
Brief Title: Stand-alone Totally Thoracoscopic Left Atrial Appendage Occlusion Using AtriClip® Device in Non-valvular Atrial Fibrillation.
Acronym: THORACS-LAAO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland (Other)
Responsible Party: Principal Investigator, Piotr Suwalski, PhD, Doctor of Philosophy, Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland
Other Study IDs: ThR-LAAO-PL
Record Dates: First submitted 2019-01-27; First posted 2019-02-12 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Stroke Prevention; Atrial Fibrillation; Safety Issues
Keywords: Stroke prevention; Atrial fibrillation; Totally thoracoscopic; LAAO; AtriClip®
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Included: The consecutive patients with atrial fibrillation assigned to totally thoracoscopic stand-alone left atrial appendage occlusion using AtriClip® for stroke prevention.
  Interventions: Device: AtriClip™ LAA Exclusion System; Drug: Oral anticoagulation therapy

INTERVENTIONS:
Device: AtriClip™ LAA Exclusion System — The left atrial appendage is closed from the epicardial side of the heart. Operative access is totally thoracoscopic. The designed and dedicated clip - AtriClip® (AtriCure, Ohio, USA) is introduced to the left pleura through thoracoscopic port.
  Other Names: AtriClip LAA Exclusion System and Delivery System (LAAØ); AtriClip LAA Exclusion System and Delivery System (PRO1); AtriClip LAA Exclusion System and Delivery System (PRO2)
Drug: Oral anticoagulation therapy — Anticoagulation therapy discontinuation - according to the standard of care at the discretion of the Investigator.

SUMMARY:
Polish multicenter registry to assess safety and durability of totally thoracoscopic left atrial appendage occlusion for stroke prevention in atrial fibrillation.

DETAILED DESCRIPTION:
The THORACS-LAAO Registry is the Polish multi-institutional registry of the consecutive patients with atrial fibrillation assigned for the totally thoracoscopic left atrial appendage occlusion (LAAO) for stroke prevention with designed epicardial clip AtriClip®. The registry has no limit of the number of patient included. Patients will be followed up with transoesophageal echocardiography at 6-12 months to assess the durability of left atrial appendage (LAA) oclusion and collect the informations about possible adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Lone atrial fibrillation
* Previous stroke or systemic thromboembolic complications
* High risk of thromboembolic complications assessed with CHA2DS2-VASc Score >2
* High bleeding risk assessed with HASBLED score => 2.
* Contraindications to oral anticoagulation
* Complications of the oral anticoagulation
* Acceptable surgical candidate, including use of general anaesthesia

Exclusion Criteria:

* Patient refusal
* Significant valve disease or coronary multi-vessel artery lesions requiring surgery
* Stroke/cerebrovascular accident (CVA) within previous 30 days
* Critical preoperative state

Intra-Operative Exclusion Criteria

* Presence of thrombus in the left atrium or LAA as documented on intra-operative transesophageal echocardiography
* LAA tissue with significant adhesions (as evaluated by the surgeon) carries AtriClip placement overly risky.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry will include all patients with atrial fibrillation with high risk of thromboembolic complications - CHA2DS2-VASc Score >2 and HASBLED score of => 2 refered to primary or secondary stroke prevention who do not require open chest surgery for other reasons.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-06-08 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Perioperative complications | First 5 postoperative days
  Number of perioperative complications associated with AtriClip placement
Intraoperative success of exclusion of LAA. | Intraoperatively
  Successful exclusion of LAA is defined as no communication between LAA and LA and < 5 mm LAA remnant measured by intraoperative transesophageal echo with Doppler.

SECONDARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCE) | 5 years
  Number of Participants with combined end point of death, acute heart failure, myocardial infarction and stroke.
Pulmonary complications. | Up to 30 days post operation
  Number of participants requiring prolonged mechanical ventilation postoperatively
Any complications connected with surgical intervention | Up to 30 days post operation
  Rate of bleeding requiring transfusion or re-operation, phrenic nerve palsy, oedema requiring intervention, wound infection, abscess in pleura

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Suwalski, PhD, Principal Investigator — Central Clinical Hospital of Ministry of the Interior and Administration in Warsaw
Locations (1):
- Central Clinical Hospital of Ministry of the Interior and Administration in Warsaw, Warsaw, Poland